CLINICAL TRIAL: NCT05986448
Title: Effects of Tai Chi for Early Pulmonary Rehabilitation in Elderly Patients With Acute Exacerbation of Chronic Obstructive Pulmonary Disease (AECOPD) and Malnutrition: a Multicenter Randomized Controlled Trial
Brief Title: Effects of Tai Chi for Early Pulmonary Rehabilitation in Elderly Patients With AECOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Houmei SHEN (Other)
Responsible Party: Sponsor-Investigator, Houmei SHEN, Senior nursing officer, Department of Emergency Medicine, Anqing Hospital Affiliated to Anhui Medical University, China, Anhui Medical University
Organization: Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-35
Record Dates: First submitted 2023-07-22; First posted 2023-08-14 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Aquatic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai-chi group (Experimental): Basic care measures and Tai-chi exercise
  Interventions: Behavioral: Tai-chi exercise
- control group (No Intervention): Basic care measures

INTERVENTIONS:
Behavioral: Tai-chi exercise — Traditional Chinese Tai Chi Movement
  Arms: Tai-chi group

SUMMARY:
The goal of this clinical trial is to learn about the therapeutic effect of Chinese traditional exercise Tai Chi in elderly acute exacerbation of chronic obstructive pulmonary disease (AECOPD) with malnutrition. The main questions it aims to answer are:

1. Improvement of pulmonary function in patients with Tai Chi exercise;
2. Improvement of pulmonary function in patients with Tai Chi exercise.

The patients in control group were given routine nursing care model, including:

1. Providing basic nursing care and protection for patients according to their needs, paying attention to the care of patients' airways, and providing relevant protection and auxiliary interventions according to the needs of patients when carrying out nebulized inhalation interventions;
2. Customized nutritional supplementation recipes by specialists in clinical nutrition, giving high-protein and low-carbohydrate diets, and giving enteral or parenteral nutritional support to those who have insufficient food intake through the mouth;
3. Carrying out health education and psychological care to alleviate the patients' psychological burdens.

On the basis of the routine care model of the control group, a Tai Chi training program was developed in Tai Chi group. Tai Chi training lasted for a total of 6 months, with 4 training sessions scheduled per week, each session lasting about 40 minutes. Experts from Anqing Tai Chi Association were invited to guide the training. The training program consists of a 5-minute pre-training warm-up, a 30-minute Tai Chi exercise, and a 5-minute post-training stretching session. The Tai Chi training was done at a moderate intensity, with the heart rate limited to 60%~80% of the maximal heart rate, where:

maximal heart rate=220-age. Accelerometers were worn for each member to record heart rate changes during training, and when the heart rate exceeded the standard range, the exercise intensity could be adjusted to keep the heart rate within a reasonable range.

ELIGIBILITY:
Inclusion Criteria:

1. ≥60 and ≤85 years of age;
2. Clinical diagnosis of COPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria;
3. Patients admitted to the hospital for treatment of chronic, repetitive coughing and severe dyspnea;
4. NRS-2002 Nutritional Risk Screening Scale score ≧3, suggesting malnutrition;
5. Conscious, able to perform normal verbal communication and without motor dysfunction

Exclusion Criteria:

1. People with impaired consciousness or invasive mechanical ventilation who were unable to fully understand and cooperate with the experiment;
2. People with active tuberculosis, lung cancer, asthma and other diseases limiting ventilation;
3. People with impaired motor function;
4. People with serious life-threatening diseases of other systems and malignant tumors;
5. People with heart failure (NYHA stage IV).

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
BODE index | Measurements of BODE index will be taken prior to the start of the trial and at 6 months after the start of the trial.
  Body Mass Index (B), the degree of airflow obstruction (O), dyspnea (D), exercise capacity (E)
Plasma total protein | Measurements of plasma total protein will be taken prior to the start of the trial and at 6 months after the start of the trial.

SECONDARY OUTCOMES:
Plasma albumin | Measurements of plasma albumin will be taken prior to the start of the trial and at 6 months after the start of the trial.
Plasma prealbumin | Measurements of plasma prealbumin will be taken prior to the start of the trial and at 6 months after the start of the trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Anqing Hospital Affiliated to Anhui Medical University, Anqing, Anhui, China